CLINICAL TRIAL: NCT05988333
Title: The Efficacy of Psychoeducational Family Intervention for Individuals With Major Depression: a Randomized Controlled Trial
Brief Title: Psychoeducational Intervention for Families With a Member Affected by Major Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Università degli Studi di Brescia (Other); University of Bologna (Other); University of Catanzaro (Other); Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other); University of Cagliari (Other); University of Florence (Other); Università degli Studi di Ferrara (Other); University of Foggia (Other); Universita degli Studi di Genova (Other); University of Milan (Other); University of Modena and Reggio Emilia (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); University of Parma (Other); University Of Perugia (Other); University of Pisa (Other); Università Politecnica delle Marche (Other); University of Roma La Sapienza (Other); University of Rome Tor Vergata (Other); Catholic University of the Sacred Heart (Other); Università degli Studi di Sassari (Other); University of Siena (Other); Università degli studi di Trieste (Unknown); Universita di Verona (Other)
Responsible Party: Principal Investigator, Mario Luciano, Doctor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0012764/2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder, Major
Keywords: depression; caregiver; family; psychoeducation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducational Family Intervention (Experimental): The experimental intervention will be administered individually to each recruited family. Sessions will take place three times a month for a period ranging from 4 to 6 months (about 18 sessions in total). The number of sessions, as well as the frequency, may vary depending on the patient's clinical situation. Sessions will have an average duration of 60-90 minutes.
  Interventions: Other: Psychoeducational Family Intervention
- Informative intervention (Active Comparator): The informative intervention consists of five sessions, administered every 7-10 days.
  Interventions: Other: Informative intervention

INTERVENTIONS:
Other: Psychoeducational Family Intervention — Supportive intervention administered to families with a member affected by MDD
  Arms: Psychoeducational Family Intervention
Other: Informative intervention — Informative intervention administered to families with a member affected by MDD
  Arms: Informative intervention

SUMMARY:
Major depressive disorder (MDD) is the most common mental disorder. It can be a huge burden not only for the person affected by it, but also for his/her whole family. The goal of this clinical trial is to test the efficacy of a family supportive intervention called psychoeducational family intervention (PFI) compared to a brief informative intervention in families with a member affected by MDD. Families will participate in one of the two interventions for a period of 6 months more or less, and they will be asked to answer some questionnaires about how much MDD impacts on their everyday life and the patient's symptoms, in order to understand whether a more structured intervention such as PFI can be useful for families in order to better deal with this complicated illness.

DETAILED DESCRIPTION:
The present paper is a no-profit, not-funded, national, multicentric, randomized-controlled trial with blinded outcome assessments, carried out in 24 Italian University outpatient units and coordinated by the Department of Mental and Physical Health and Preventive Medicine of the University of Campania Luigi Vanvitelli. In each center, 8 patients (and their families) and 8 controls will be recruited, for a total of 192 families assigned to the experimental group and 192 to the control group (total sample size = 384 families). Families are assessed at the baseline and 6-, 12- and 24-months post-randomization.

The primary aim of this study is to assess the efficacy of PFI in a group of patients with a diagnosis of MDD in terms of: 1) reduction of depressive symptoms; 2) improvement of psychosocial functioning; 3) improvement of social network. Furthermore, the efficacy of PFI will be also evaluated in terms of: 1) reduction of relapses and hospitalization in the 18 months following the end of the intervention; 2) improvement of adherence to pharmacological treatments and of patients' quality of life; 3) reduction of self-stigma; 4) improvement of coping strategies, family burden, and expressed emotion of family members of patients with major depression; 5) improvement of quality of life of family members. Finally, our study will investigate whether the presence of specific temperamental profiles and childhood traumas may mediate the effectiveness of the psychoeducational intervention.

The experimental intervention consists of the psychoeducational family intervention developed by Ian Falloon for the treatment of schizophrenia, which has been adapted to major depression and to the Italian context. The experimental intervention will be administered individually to each recruited family and consists of six phases: 1) engagement of the family unit; 2) individual assessment; 3) family assessment; 4) informative sessions; 5) communication skills sessions; 6) problem-solving skills sessions.

Patients and their relatives will be provided with information on: 1) the clinical characteristics of MDD, including onset and course, symptoms, prognosis, risk and protective factors; 2) available pharmacological and non-pharmacological treatments of MDD, its indications, side effects and strategies to cope with them, treatment duration, risk factors for relapse, and effects related to abrupt cessation of the therapy; 3) early signs of crisis, with the identification of the user's specific signs, completion and use of an ad-hoc form, the usefulness of their recognition for the prevention of episodes. A specific informative session on suicide has been developed, which will be administered only if the patients had a previous suicide attempt or report suicidal ideation during the intervention.

Each meeting is ideally divided into three phases: a first phase dedicated to clarifications and questions regarding the topics previously discussed; a second phase focused on the main topic of the meeting (the so-called "teaching phase"); and a final phase, in which the salient aspects discussed during the meeting are summarized, and "homework" is assigned.

The control group will receive an informative intervention consisting of five sessions, administered every 7-10 days, with the following content: healthy lifestyle habits (diet and nutrition), stress management, regulation of circadian rhythms, and management of medications' side effects.

The interventions will be discontinued if: 1) patients or their relatives will be unable to attend more than five consecutive psychoeducational sessions; 2) patients will be hospitalized or had any affective relapse during the intervention; or 3) patients or relatives withdraw their consent.

In both groups, patients will continue to receive the treatment usually provided in their center.

Trainings for the conduction of the intervention and for the use of assessment tools will be provided by the coordinating center. Two researchers (at least one being a psychiatrist) for each center will participate in a four-day training. During the training, a manual to conduct the experimental intervention is provided to participants, and several role-plays are organized. At least one researcher per center, not involved in the administration of the interventions, will be trained in the use of assessment tools and inter-rater reliability measurement. The training will include the following phases: a) presentation of the assessment instruments; b) group reading; c) simulations of administration; d) video-recorded interviews.

Work hypotheses is that the PFI will be effective in reducing severity of depressive symptoms, relapses and hospitalizations, and an improvement in adherence to pharmacological treatments, quality of life a reduction in internalized stigma, and an improvement in coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of major depression, according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition;
* ability to provide informed consent;
* presence of at least one contact per month with the psychiatric clinic for at least six months prior to recruitment;
* cohabitation with at least one family member.

Exclusion Criteria:

* moderate or severe cognitive deficits, physical illnesses preventing the participation to the sessions or if they were hospitalization in the two months prior the enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Severity of depressive symptoms | At baseline, after 6-, 12- and 24 months
  Hamilton Depression Rating Scale (HAM-D). The HAM-D includes 17 items. Of these, 8 items are scored from 0 (absent) to 4 (severe), while nine are scored from 0 to 2. The total score is performed by the sum of the items' scores, and ranges from 0 to 52 points.
Psychosocial functioning | At baseline, after 6-, 12- and 24 months
  Personal and Social Performance Scale (PSP). A total score can be attributed to score the overall patient's functioning, ranging from 0 to 100, with higher scores indicating higher functioning. Ratings are based mainly on the assessment of patient's functioning in four main areas: (1) socially useful activities; (2) personal and social relationships; (3) self-care; and (4) disturbing and aggressive behaviors.
Severity of anxiety symptoms | At baseline, after 6-, 12- and 24 months
  Hamilton Anxiety Rating Scale (HAM-A). It is a 14-items questionnaire developed to measure the severity of anxiety symptoms, both psychic (mental agitation and psychological distress) and somatic (physical complaints related to anxiety). The score for each item ranges from 0 (not present) to 4 (extreme severity).
Social contacts | At baseline, after 6-, 12- and 24 months
  Columbia Suicide Severity Rating Scale (C-SSRS). The clinician-administered version of the C-SSRS (screening version) will be administered. Individual's suicidal ideation is rated on a scale from 1 (wish to be dead) to 5 (active suicidal ideation with a specific plan and intent).
  Social Network Questionnaire (SNQ).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania L. Vanvitelli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No